CLINICAL TRIAL: NCT04913844
Title: Effect of Ski Sport on Physical Performance, Pain, Quality of Life, and Gender Differences
Brief Title: Effect of Ski Sport on Physical Performance
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Arzu Keskin Aktan, Principal Investigator, Afyonkarahisar Health Sciences University
Other Study IDs: 2018/598
Record Dates: First submitted 2021-05-27; First posted 2021-06-04 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Physical Performance; Pain; Quality of Life
Keywords: Skiing; Gender difference; Muscle strength; Physical performance; Pain; Quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Skiers group: The skiers group was formed from licensed ski athletes (17 male, 17 female) who have been active in sports for at least the last 2 years.
  There will be no interventions. Physical performance tests and observational assessments will be conducted.
  Interventions: Other: Physical performance tests and observational assessments
- Control group: The control group was composed of non-athletic and age-matched participants (17 male, 17 female) with no skiing experience.
  There will be no interventions. Physical performance tests and observational assessments will be conducted as in the Skiers Group.
  Interventions: Other: Physical performance tests and observational assessments

INTERVENTIONS:
Other: Physical performance tests and observational assessments — There will be no interventions. Physical performance tests and observational assessments will be conducted.

SUMMARY:
The aim of the study is to investigate the effect of ski sport on physical performance, pain, and quality of life compared to sedentary individuals of similar age groups and to examine the existence of gender-specific differences.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effects of skiing on physical performance, pain, quality of life, and gender-specific differences. In this context, aerobic/anaerobic performance, body balance, hand-grip strength, and back-leg-chest strength were evaluated in male and female ski athletes and age- and sex-matched sedentary controls.

In addition, pain experiences, low back pain-related disability level, and quality of life of all participants were questioned using SF 36, McGill Pain Questionnaire (MPQ), Oswestry Low Back Pain Disability Questionnaire (OLBPDQ), and VAS scales.

The data thus collected were used to determine whether skiing had any effect on physical performance and quality of life, as well as the possible impact of skiing on gender-specific differences.

ELIGIBILITY:
Inclusion Criteria:

Skiers Group;

* Being an active athlete for at least the last 2 year and affiliated with the National Ski Federation
* International Physical Activity Questionnaire-Short Form (IPAQ-SF) total score above 3000 METs min/week

Control Group;

* Being healthy and non-athletic with no ski experience
* Having similar sociodemographic characteristics with Skiers Group
* IPAQ-SF total score below 3000 METs min/week

Exclusion Criteria:

* History of surgery and/or serious trauma to the spine, lower and upper extremity,
* Chronic illnesses
* Substance addiction such as cigarette-alcohol, etc.
* During the study; the need of receiving treatment/ interventions due to trauma or any other conditions is concluded with withdrawal from the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample of the study consists of a total of 68 participants between the ages of 18-25. Licensed ski athletes in Turkey (17 male, 17 female), who have been active in sports for at least the last 2 years, were included in the skiers group, and an age-matched non-athletic person (17 male, 17 female) with no skiing experience was included in the control group. The evaluations of the Skiers group were made at Erciyes Ski Center, and those of the control group were made at the Faculty of Health Sciences of Nuh Naci Yazgan University.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | 5 minutes
  The International Physical Activity Questionnaire-Short Form (IPAQ-SF), the short form of which consists of 7 questions, is a self-reported scale that is widely used to measure physical activity level.Based on the guidelines, the IPAQ score is calculated as metabolic equivalents (METs) per minutes per week, and the IPAQ score below 3000 METs-min / week indicates a low-moderate physical activity level. Total IPAQ score <3000 METs min / week was used to determine the sedentary control group as the inclusion criteria.
The Young Men's Christian Association (YMCA) Step Test | 10 minutes
  The Young Men's Christian Association (YMCA) step test is a test that can be used in athletes and non-athletes and correlates heart rate with cardiovascular fitness level. For this test, participants are asked to climb up and down a 12-inch step for 3 minutes (metronome set at 96 beats per minute). The heart rate measurement, which is continued for 1 minute immediately after the end of the test, is recorded as beats / min. The low heart rate measured in the step tests indicates a high level of cardiovascular fitness.
Vertical Jump Test (VJT) | 10 minutes
  The Vertical Jump Test (VJT) is an effective test used to indirectly evaluate the anaerobic performance of participants. In this test, the difference in centimeters is recorded between the maximum height attainable with the arm of the participant whose dominant side stands at the edge of the wall and the maximum height attained by jumping. The measurement is repeated 3 times with rest periods and the maximum value is recorded in cm
Flamingo Balance Test (FBT) | 5 minutes
  The Flamingo Balance Test (FBT) is used to measure coordination of full body equilibrium. In the FBT, the number of errors that the participants made within 60 seconds on the flamingo balance board is recorded.
Hand-Grip Strength (HGS) | 5 minutes
  Hand-grip strength (HGS) measurement is made with a hydraulic hand-grip dynamometer. HGS measurement is performed for the dominant hand when the elbow is close to the body, 90 degrees of flexion, and the wrist is in a neutral position. The measurement is repeated 3 times and the maximum value is recorded in kg. The dominant hand is determined by asking the participants with which hand they write.
Back-Leg-Chest Strength (BLCS) | 10 minutes
  The BLC dynamometer is used to measure back-leg-chest strength (BLCS) in a single measurement. BLCS measurements are used as a suitable measure to characterize overall body strength. The measurement is repeated 3 times with rest periods and the maximum value is recorded in kg.
Visual Analog Scale (VAS) | 5 minutes
  VAS is a widely used and reliable scale for evaluating pain intensity. With VAS, the severity of pain experienced in various situations such as 1) rest, 2) activity, and 3) most severe pain experienced (MSPE) can be evaluated. In addition to this study, VAS-skiing was added only to the skiers group. Participants are asked to mark the level of pain they feel on a 10 cm straight line marked as "no pain (0)" at one end and "unbearable pain (10)" at the other end. The distance between the marked point and the starting point is measured and recorded in cm.
Short Form-36 (SF-36) Quality of Life Questionnaire | 15 minutes
  Short Form-36 (SF-36) is a valid and reliable self reported scale. SF-36 is generally used to evaluate health-related quality of life of individuals aged 14 and over. SF-36 has eight sub-dimensions such as physical functioning, role limitation by physical problems, bodily pain, general health, vitality, social functioning, role limitation by emotional problems, and mental health. Separate scores are calculated for each sub-dimension. The scores of the sub-dimensions range from 0 to 100. High scores on the scale indicate an increase in quality of life, and a low score indicates a decrease in quality of life.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire (OLBPDQ) | 10 minutes
  OLBPDQ is a valid and reliable self reported scale. OLBPDQ consists of 10 items that assess different aspects of the function, such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and changing degree of pain. In the 6-point Likert type scale, the first expression is scored as '0' and the sixth expression as '5'. The total score is multiplied by 2 and expressed as a percentage. The increase in the ODI score (Range 0--100%) indicates the increase in the level of disability and the disability level is classified as follows: 0-20% (minimal disability), 21-40% (moderate disability), 41-60% (severe disability), 61 -80% (crippled), 81-100% (patients who are either bed-ridden or exaggerate their symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Keskin Aktan, Study Director — Afyonkarahisar Health Sciences University; Nilüfer Keskin Dilbay, Principal Investigator — Marmara University; Özden Kutlay, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not plan to make IPD available.